CLINICAL TRIAL: NCT00661492
Title: A Randomized Phase II Study of Mitoxantrone vs. Mitoxantrone With Cetuximab in Metastatic Androgen Independent Prostate Cancer (AIPC) Previously Treated With Docetaxel-based Chemotherapy
Brief Title: Mitoxantrone ± Cetuximab 2nd Line Androgen Independent Prostate Cancer (AIPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Eli Lilly and Company (Industry); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-118
Record Dates: First submitted 2008-04-04; First posted 2008-04-18 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Androgen-independent Prostate Cancer
Keywords: Androgen-independent prostate cancer(AIPC)
MeSH Terms: interventions — Cetuximab; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Erbitux (cetuximab) and Novantrone (mitoxantrone)
  Interventions: Drug: cetuximab; Drug: Mitoxantrone
- Arm 2 (Experimental): Novantrone (mitoxantrone)
  Interventions: Drug: Mitoxantrone

INTERVENTIONS:
Drug: cetuximab — Erbitux (cetuximab) IV over 2 hours (loading dose) on Day 1 (Cycle 1 only), followed by Erbitux (cetuximab) IV over 1 hour weekly thereafter
  Other Names: Erbitux
  Arms: Arm 1
Drug: Mitoxantrone — Novantrone (mitoxantrone) IV Day 1 + Prednisone QD for ten (10) 21-day cycles Standard androgen deprivation therapy (ADT) will be continued in all patients who enter study on LHRH agonists
  Other Names: Novantrone

SUMMARY:
To determine the time to progression produced by the combination of Novantrone (mitoxantrone) and Erbitux (cetuximab) versus Novantrone alone in metastatic AIPC patients previously treated with docetaxel-based chemotherapy. TTP is defined as time from the start of treatment date to the date the patient is first recorded as having disease progression, even in patients who discontinue study treatment early due to toxicity.

DETAILED DESCRIPTION:
This is a nonblinded, randomized phase II study to determine the activity of Novantrone (mitoxantrone) with or without Erbitux (cetuximab) in patients with androgen independent prostate cancer (AIPC) who have been treated previously with docetaxel chemotherapy. The Novantrone (mitoxantrone)-only treatment arm will serve as a concurrent control arm to aid in the determination of the benefit of the Novantrone (mitoxantrone)-Erbitux (cetuximab) combination in this setting.

Patients will be randomly assigned 2:1 to 1 of 2 treatment arms; 93 patients in Arm 1 and 47 patients in Arm 2. A balanced randomization procedure will be performed utilizing a code list that will be developed prior to the study opening. Because the patients will be stratified by performance status (ECOG 0 and 1 vs. ECOG 2), the list will be developed to ensure a balance between the 2 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate. Note: Patients may have either measurable or non-measurable disease.
* Radiographic evidence of regional or distant metastases
* Current evidence of progression (by PSA and/or imaging studies) despite standard hormonal therapy.
* Progression by PSA will be defined as: A rising PSA defined as: at least 2 rises in PSA over a reference value (PSA #1). The first rising PSA (PSA #2) must be taken at least 1 week after PSA #1. A third PSA (PSA #3) is required to be greater than PSA #2; if not, a fourth PSA (PSA #4) is required to be greater than PSA #2. Progression for nonmeasurable disease will be defined as 2 or more new bone lesions; for measurable disease, progression will be defined by standard RECIST criteria.
* For patients who have been on antiandrogen therapy (ie, bicalutamide, flutamide, etc.), patients must have discontinued anti-androgen therapy for at least 6 weeks (4 weeks for flutamide) without evidence of an antiandrogen withdrawal response. A washout period will not be required for patients who did not respond to an antiandrogen prescribed as second line hormonal therapy. For patients whose progression is documented by PSA, the last required PSA must be after the required anti-androgen washout period (4-6 weeks as appropriate).
* One prior docetaxel-containing regimen. Patients must have received at least 2 doses in an every 3-week schedule or 6 doses on a weekly schedule of docetaxel. Patients may have discontinued therapy due to progression, intolerance, completion of planned therapy, or other reasons. Chemotherapy treatment with any second-line regimen will not be permitted. Patients who have been previously treated with a first-line docetaxel-based doublet regimen will be eligible for this study, (eg, patients treated on a prior first-line trial containing a docetaxel/carboplatin or other docetaxel-based doublet).
* Serum testosterone levels (See protocol for specific details) (unless surgically castrate). Patients must continue androgen deprivation with an LHRH agonist if they have not undergone orchiectomy
* ECOG performance status
* Laboratory criteria for entry:

  * absolute neutrophil count
  * platelets
  * bilirubin
  * AST or ALT
* Life expectancy greater than 3 months
* Age greater than or equal to 18 years
* Agree to use contraceptives while on study if sexually active, and for 2 months after the last dose of study drug.
* Has signed a Patient Informed Consent Form
* Has signed a Patient Authorization Form

Exclusion Criteria:

* More than 1 prior chemotherapy regimen for metastatic disease
* Prior history of uncontrolled congestive heart failure or left ventricular ejection fraction (LVEF) that is less than the institution's lower limit of normal on MUGA or echocardiogram
* A second active malignancy (diagnosed within 5 years) except adequately treated non-melanoma skin cancer or other non-invasive or in-situ neoplasm
* Significant active concurrent medical illness or infection
* Treatment with chemotherapy for AIPC within the past 21 days
* Prior treatment with Novantrone (mitoxantrone)
* Prior therapy which specifically and directly targets the EGFR pathway
* Prior severe infusion reaction to a monoclonal antibody
* Recent myocardial infarction (within prior 6 months)
* Prior treatment with radionuclides, with the exception of prior treatment with samarium, which will be allowed provided at least 8 weeks have passed since administration.
* Is receiving concurrent immunotherapy, hormonal therapy, radiation therapy, or any other non-protocol therapy (excluding LHRH antagonist)
* Is receiving concurrent investigational therapy or has received such therapy within the past 30 days
* Has evidence of CNS involvement
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection.
* Is unable to comply with requirements of study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark T. Fleming, MD, Principal Investigator — Virginia Oncology Associates/US Oncology
Locations (54):
- United States (54):
  - Hematology Oncology Associates, Phoenix, Arizona
  - Northern AZ Hematology & Oncology Assoc, Sedona, Arizona
  - Rocky Mountain Cancer Center-Midtown, Denver, Colorado
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Florida Cancer Institute - New Hope, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Hope Center, Terre Haute, Indiana
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - NH Oncology-Hematology PA, Hooksett, New Hampshire
  - Hematology-Oncology Associates of NNJ, P, Morristown, New Jersey
  - Albany Medical Cancer Center, Albany, New York
  - Interlakes Oncology Hematology, PC, Rochester, New York
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Oncology, P.A. -Amarillo, Amarillo, Texas
  - Texas Oncology, P.A., Arlington, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Methodist Charlton Cancer Ctr., Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Texas Oncology, P.A, Garland, Texas
  - Longview Cancer Center, Longview, Texas
  - South Texas Cancer Center - McAllen, McAllen, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - Texas Oncology - Odessa, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology Cancer Center-Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology, P.A., Webster, Texas
  - Fairfax Northern VA Hem-Onc PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onc and Hem Associates of SW VA, Inc., Salem, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Puget Sound Cancer Center-Edmonds, Edmonds, Washington
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
  - Puget Sound Cancer Center-Seattle, Seattle, Washington
  - Cancer Care Northwest-South, Spokane, Washington
  - Northwest Cancer Specialists-Vancouver, Vancouver, Washington
  - Yakima Valley Mem Hosp/North Star Lodge, Yakima, Washington

REFERENCES:
- [Derived] Fleming MT, Sonpavde G, Kolodziej M, Awasthi S, Hutson TE, Martincic D, Rastogi A, Rousey SR, Weinstein RE, Galsky MD, Berry WR, Wang Y, Boehm KA, Asmar L, Rauch MA, Beer TM. Association of rash with outcomes in a randomized phase II trial evaluating cetuximab in combination with mitoxantrone plus prednisone after docetaxel for metastatic castration-resistant prostate cancer. Clin Genitourin Cancer. 2012 Mar;10(1):6-14. doi: 10.1016/j.clgc.2011.11.003. PMID 22340631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2008 and March 2009, 115 eligible patients were enrolled, 75 in the CMP arm and 40 in the MP arm.
Pre-assignment Details: 5 patients with Withdrew Consent and 23 patients with Failed Entry.
Groups:
- Arm 1: Novantrone+Erbitux
- Arm 2: Novantrone
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 75 | 40
Completed | 7 | 11
Not Completed | 68 | 29
Not completed — Adverse Event | 16 | 13
Not completed — Disease Progression | 44 | 14
Not completed — Patient Request | 6 | 1
Not completed — Investigator Request | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 75 | 40 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 8 | 25
  >=65 years | 58 | 32 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (8.7) | 70.7 (8.1) | 71.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 75 | 40 | 115
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 65 | 32 | 97
  Hispanic | 4 | 3 | 7
  Black | 5 | 5 | 10
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 75 | 40 | 115

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression (TTP)
Description: TTP will be measured from the start of treatment date to the date the patient is first recorded as having disease progression (even in patients who discontinue study treatment early due to toxicity or death due to disease progression.
Time Frame: 24 months
Population: ITT population
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 75 | 40
Months | 4.9 [0.5 to 20.5] | 6.6 [0.3 to 23.1]

2. Secondary Outcome: 2-year Radiographically Evident Progression-free Survival (REPFS).
Description: Radiographic progression:
  1) For bone scan, 2 unequivocal new lesions confirmed by a subsequent bone scan with at least 1 more new lesion; 2) Skeletal related event (eg, fracture, need for radiation to bone for pain, spinal cord compression, need for surgery to bone to prevent or treat a pathologic fracture).
Time Frame: 24 months.
Population: Patients who received bone scans or had bone progression only (bone pain/pathologic fracture/palliative radiation).
Measure: Number (95% Confidence Interval); unit: Probability of REPFS at 2-year
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 50 | 24
Probability of REPFS at 2-year | 0.73 [0.56 to 0.85] | 0.80 [0.55 to 0.92]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR = CR + PR Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: 24 months
Population: Patients with solid tumors
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 45 | 26
percentage of participants | 2.2 [0.1 to 11.8] | 3.8 [0.1 to 19.6]

4. Secondary Outcome: Median Time to Prostate-specific Antigen (PSA) Progression
Description: Defined as the time from initiation of therapy until the first 25% increase from baseline in non-responders or 50% increase from nadir in responders as defined above. A minimum increase in the PSA of 5 ng/mL will be required for progression.
Time Frame: 24 months
Population: Patients with Prostate-specific antigen (PSA) Information
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 65 | 34
Months | 2.7 [0.03 to 24.1] | 2.7 [0.03 to 22.3]

5. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate
Description: Defined as the fraction of patients with a ≥50% reduction in serum PSA confirmed by a second serum PSA at least 3 weeks later
Time Frame: 24 months
Population: Evaluable Population with Prostate-specific antigen (PSA) Information
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 65 | 34
percentage of participants | 7.7 [2.5 to 17.0] | 17.6 [6.8 to 34.5]

6. Secondary Outcome: Prostate-specific Antigen (PSA) Doubling Time
Description: PSA doubling time = [log (2)× t] ÷ [log (final PSA) - log (initial PSA)]
Time Frame: 24 months
Population: Evaluable Population with Prostate-specific antigen (PSA) Information
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 65 | 34
months | 2.3 [-61.3 to 62.8] | 1.5 [-2544 to 76.4]

7. Secondary Outcome: Median Progression-free Survival (PFS)
Description: PFS is measured from the date of randomization to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at last contact date.
Time Frame: 24 months
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 75 | 40
months | 4.2 [0.5 to 20.5] | 5.5 [0.3 to 23.1]

8. Secondary Outcome: Median Overall Survival (OS)
Description: OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: 30 months
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 75 | 40
months | 11.9 [0.5 to 24.1] | 15.7 [0.9 to 29.4]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose
Description: For treated patients only, assessed at each treatment visit
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 39/75 | 12/39
Other Adverse Events (participants affected / at risk) | 74/75 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=75) | Arm 2 (N=39)
ACCIDENT CEREBROVASCULAR (Vascular disorders) | 0 (0) | 1 (1)
ALLERGIC REACTION (Immune system disorders) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
ANOREXIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
BELL'S PALSY (Nervous system disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Vascular disorders) | 1 (1) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0)
CONFUSION (Nervous system disorders) | 1 (1) | 0 (0)
CONGESTIVE HEART FAILURE (Vascular disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 3 (3) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DISTRESS RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 1 (1)
EDEMA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
EFFUSION PLEURAL (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
EMBOLISM PULMONARY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
EMBOLUS PULMONARY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEVER (Infections and infestations) | 1 (1) | 0 (0)
BRAIN METASTASES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DEATH SUDDEN (NOS) (Investigations) | 1 (1) | 0 (0)
DISEASE PROGRESSION (Investigations) | 4 (4) | 0 (0)
FIBRILLATION ATRIAL (Cardiac disorders) | 1 (1) | 1 (1)
FLUTTER ATRIAL (Cardiac disorders) | 1 (1) | 0 (0)
FRACTURE PATHOLOGICAL (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI HEMORRHAGE (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 1 (1) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
INFECTION BACTERIAL (Infections and infestations) | 4 (4) | 0 (0)
INFECTION BLADDER (Infections and infestations) | 3 (3) | 0 (0)
INFECTION VIRAL (Infections and infestations) | 1 (1) | 0 (0)
ISCHEMIA MYOCARDIAL (Cardiac disorders) | 1 (1) | 0 (0)
MENTAL DEFICIENCY (Nervous system disorders) | 1 (1) | 0 (0)
MENTAL DETERIORATION (Nervous system disorders) | 0 (0) | 1 (1)
MOOD ALTERED (Psychiatric disorders) | 0 (0) | 1 (1)
MULTIPLE ORGAN FAILURE (General disorders) | 1 (1) | 0 (0)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
NOSEBLEED (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 2 (2) | 0 (0)
PAIN BACK (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PAIN PELVIC (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
PAIN SACROILIAC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PHLEBITIS (Vascular disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
PROSTATIC DISORDER (Endocrine disorders) | 1 (1) | 0 (0)
RECTAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 1 (1)
RECTAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Gastrointestinal disorders) | 3 (3) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
SPINAL CORD COMPRESSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
STROKE (Vascular disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (2) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 1 (1) | 2 (2)
TRACHEOBRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
URINARY BLADDER OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
WEAKNESS (General disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=75) | Arm 2 (N=39)
NEUTROPENIA (Blood and lymphatic system disorders) | 48 (139) | 14 (35)
FATIGUE (General disorders) | 36 (50) | 22 (34)
LEUCOPENIA (Blood and lymphatic system disorders) | 27 (141) | 10 (23)
RASH (Skin and subcutaneous tissue disorders) | 25 (63) | 3 (3)
ANEMIA (Blood and lymphatic system disorders) | 24 (50) | 15 (41)
PAIN (General disorders) | 24 (35) | 12 (17)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 23 (58) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 17 (29) | 11 (13)
ANOREXIA (Gastrointestinal disorders) | 17 (19) | 10 (11)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 17 (56) | 8 (14)
DRY SKIN (Skin and subcutaneous tissue disorders) | 17 (26) | 4 (4)
CONSTIPATION (Gastrointestinal disorders) | 16 (20) | 9 (9)
DIARRHEA (Gastrointestinal disorders) | 14 (22) | 9 (10)
EDEMA (Blood and lymphatic system disorders) | 13 (15) | 7 (8)
VOMITING (Gastrointestinal disorders) | 12 (19) | 9 (10)
DIZZINESS (Nervous system disorders) | 12 (18) | 7 (9)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 11 (19) | 6 (9)
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 4 (4)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 4 (5)
INFECTION BACTERIAL (Infections and infestations) | 10 (13) | 1 (1)
PAIN BACK (Musculoskeletal and connective tissue disorders) | 9 (13) | 6 (8)
MUCOSITIS (Gastrointestinal disorders) | 9 (14) | 4 (4)
WEAKNESS (General disorders) | 9 (10) | 3 (3)
FEVER (Infections and infestations) | 9 (10) | 2 (2)
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 7 (11) | 4 (4)
ALLERGIC REACTION (Immune system disorders) | 7 (8) | 2 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 6 (15) | 9 (19)
INFECTION UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
INSOMNIA (Nervous system disorders) | 6 (6) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 (9) | 2 (2)
WEIGHT LOSS (General disorders) | 6 (6) | 2 (2)
HEADACHE (Nervous system disorders) | 5 (5) | 5 (5)
DEHYDRATION (Gastrointestinal disorders) | 5 (9) | 4 (4)
NEUROPATHY (Nervous system disorders) | 5 (5) | 3 (3)
HEMATURIA (Renal and urinary disorders) | 5 (6) | 2 (3)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
CHILLS (General disorders) | 5 (5) | 1 (3)
CONJUNCTIVITIS (Eye disorders) | 5 (6) | 1 (1)
INFECTION FUNGAL (Infections and infestations) | 5 (9) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 5 (37) | 1 (1)
MUSCLE WEAKNESS (General disorders) | 5 (9) | 1 (1)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 5 (5)
ALKALINE PHOSPHASTASE SERUM INCREASE (Metabolism and nutrition disorders) | 4 (4) | 4 (8)
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
INFECTION BLADDER (Infections and infestations) | 4 (6) | 3 (3)
CELLULITIS (Infections and infestations) | 4 (7) | 2 (2)
URINARY URGENCY/FREQUENCY (Renal and urinary disorders) | 4 (4) | 1 (1)
ANXIETY (Psychiatric disorders) | 4 (4) | 0 (0)
CHEST PAIN (General disorders) | 4 (4) | 0 (0)
EPIPHORA (Eye disorders) | 4 (4) | 0 (0)
GLUCOSE BLOOD INCREASED (Metabolism and nutrition disorders) | 4 (8) | 0 (0)
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
ALT INCREASED (Metabolism and nutrition disorders) | 3 (5) | 2 (6)
AST INCREASED (Metabolism and nutrition disorders) | 3 (7) | 2 (4)
CREATININE SERUM INCREASED (Metabolism and nutrition disorders) | 3 (9) | 2 (3)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
HYPOTENSION (Vascular disorders) | 2 (3) | 2 (2)
THROMBOSIS (Vascular disorders) | 2 (2) | 2 (2)
CARDIAC INSUFFICIENCY (Cardiac disorders) | 1 (1) | 4 (4)
DYSGUESIA (Gastrointestinal disorders) | 1 (1) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 2 (2)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
RECTAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 2 (3)
BRUISE (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No